CLINICAL TRIAL: NCT06546826
Title: Alveolar Ridge Preservation With Several Techniques: a Multicenter Observational Longitudinal Study
Brief Title: Alveolar Ridge Preservation After Tooth Extraction
Acronym: CRES-PRES
Status: Active, not recruiting | Type: Observational
Sponsor: International Piezosurgery Academy (Other)
Collaborators: Universidade do Porto (Other); University of Trieste (Other)
Responsible Party: Principal Investigator, Mr. Claudio Stacchi, DDS, MSc, Head of Scientific committe of International Piezosurgery Academy, International Piezosurgery Academy
Other Study IDs: 207_2022
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Alveolar Bone Loss
Keywords: tooth extraction; implant insertion; post extraction bone remodeling
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — alveolar bone specimens withdrawn with trephine bur
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- BARP: collagen-bonegraft-collagen
  Interventions: Procedure: BARP
- unassisted: unassisted healing
  Interventions: Procedure: simple tooth extraction
- Tooth root: tooth root and PRF
  Interventions: Procedure: tooth root and PRF
- Ice Cream Cone Technique: bonegraft and collagen membrane

INTERVENTIONS:
Procedure: BARP — deep layers of collagen, medium-superficial heterologous bone graft, superficial collagen layer
  Other Names: Biologically-oriented Alveolar Ridge Preservation
  Groups: BARP
Procedure: simple tooth extraction — tooth extraction without grafting procedure.
  Groups: unassisted
Procedure: tooth root and PRF — Autogenous roots derived from the extracted hopeless tooth and stabilized with osteosynthesis screws to reconstruct the missing buccal wall of the socket. The defect was then filled with PRF.
  Groups: Tooth root
Procedure: Ice cream cone technique — xenogeneic granules and a resorbable collagen membrane

SUMMARY:
Post-extractive alveolar ridge remodeling represents a physiological phenomenon that may hamper successive implant insertion. Several techniques have been proposed without any significant difference of efficacy among them. Moreover several research protocols of analysis have been proposed, including histomorphometric, radiological, clinical analysis.

The purpose of the present study is to test different alveolar ridge preservation techniques using histomorphometric and optical scanning analysis.

DETAILED DESCRIPTION:
Primary objective The primary objective of the study is to clinically compare the effect on the preservation of the alveolar ridge using different techniques (dental roots in association with platelet rich fibrin, BARP (Biologically-oriented Alveolar Ridge Preservation), Ice Cream Cone Technique and unassisted socket healing).

Secondary objective The secondary objective is the collection of histological and histomorphometric data that allow to evaluate the quality and quantity of newly formed bone.

Study design Multicenter observational study of a prospective non-profit case-control.

List of centers involved in addition to our facility:

- University of Porto, Faculty of Dentistry, Specialization in Periodontology and Implantology.

Study population The study will be conducted in an outpatient hospital setting.

Number of patients to be enrolled to compare autogenous tooth roots (TR) and ice cream cone technique (ICCT): 32 patients among all the centers involved, of which 16 patients in the University of Porto and 16 patients in University of Trieste center including dropouts.

Number of patients to be enrolled to compare BARP and unassisted socket healing: 30 patients in the University of Trieste including dropouts.

Enrollment procedure All patients who meet the inclusion and exclusion criteria will be enrolled in the study following the administration of the Information Sheet and the acquisition of informed consent.

The choice of the alveolar ridge preservation protocol will be motivated by the clinicians experience and the patients preference among those currently validated (ice-cream cone technique, tooth root, etc.).

Autogenous tooth roots: under local anesthesia, a trapezoidal mucoperiosteal flap, extended to adjacent teeth mesially and distally, will be raised to expose the defect and remove granulation tissue. The dental root graft will be obtained by sectioning the extracted tooth at the cementoenamel junction and then separating the root longitudinally to fully expose the pulp chamber using a tungsten carbide bur with irrigation. The specimen will then be thoroughly cleaned using manual curettes on the external surface, while the removal of residual pulp tissue and/or root canal filling material will be performed using a tungsten carbide bur with irrigation. The tooth root specimen will be resized to fit the height and width of the post-extraction site to be regenerated and fixed using one to two titanium osteosynthesis screws. A blood sample will then be collected in two sterile glass-lined plastic tubes and processed to produce a platelet rich fibrin membrane. The blood sample will be centrifuged (2700 rpm for 12 minutes). The platelet rich fibrin will then be removed from the tubes and placed on the surgical site. Periosteal releasing incisions will be made to advance the mucoperiosteal flap, which will be repositioned coronally and secured with horizontal mattress sutures and single stitches to ensure a submerged healing condition.

Ice Cream Cone technique: under local anesthesia, the compromised tooth will be extracted atraumatically without raising a flap. A resorbable collagen membrane will be shaped into a cone and inserted into the socket, into which the xenograft will be placed; mattress sutures will then be placed.

BARP: under local anesthesia, the compromised tooth will be extracted atraumatically without raising a flap. After granulation tissue removal, the socket will be filled with a collagen sponge (deep collagen layer) up to 4 to 5 mm from the most coronal extensions of the buccal crest to create a support for the intra-alveolar graft. A bovine derived xenograft will be placed on top of the collagen sponge to fill the coronal part of the socket, avoiding overfilling (graft layer). Socket sealing will be performed with a new layer of collagen sponge that will be placed over the exposed portion of the graft layer and firmly held by sutures.

For all patients, after 26 weeks of healing, a mucoperiosteal flap will be raised to expose the target site and a titanium implant will be inserted. During this phase, using a core drill to prepare the implant site, it will also be functional to obtain a bone sample that will be subsequently analyzed.

Study Outcomes

The primary endpoint is the width of the alveolar ridge, which will be assessed in two stages:

* T0: initial condition of the alveolar ridge, measured before performing surgery;
* T1: final condition of the alveolar ridge, measured before implant insertion at 26 weeks of healing from surgery.

The primary endpoint will be classified as follows. The secondary endpoints are represented by histomorphometric variables: newly formed mineralized tissue (New bone/Total volume), graft residues (RG/TV), newly formed non-mineralized tissue (Nonmineralised tissue/Total volume), total mineralized tissue that will be assessed at twenty-six weeks of healing (Mineralised tissue/total volume) evaluated as means and standard deviations and with χ2 test.

The primary endpoint will then be assessed in relation to complications and adverse events, such as:

* Soft tissue dehiscence;
* Graft exposure;
* Graft loss;
* Wound infections.

The width of the alveolar ridge will be measured linearly and volumetrically, using digital scans processed by a 3D scanning software (Geomagic Control X, 3D System, Morrisville, USA) at the University of Trieste.

The data collected at follow-up and the outcome data are based on a clinical evaluation, considering the possible presence of complications and adverse events.

The histological and histomorphometric analysis of all samples will be performed by one of the authors, blinded to the study design and the origin of the biopsy. The biopsies, left inside the core drills to maintain the orientation of the bone core, will be rinsed with a cold 5% glucose solution to remove blood residues while maintaining the correct osmolarity (278 mOsm/L). The samples will then be fixed for 3 days in a 10% buffered formalin solution at pH 7.2 and then processed for histological and histomorphometric evaluation at the Bone Lab, University of Trieste. After this, the samples will be delivered to specialized and authorized companies for disposal, according to current legislation.

Collected data variables and sources

The following variables will be collected for each enrolled patient/participant:

* Width of the alveolar ridge;
* Newly formed mineralized tissue, graft residues, non-mineralized newly formed tissue, total mineralized tissue.

Histological and histomorphometric analysis of all samples will be performed by one of the authors, blinded to the study design and biopsy origin. Biopsies, left inside the core drills to maintain the orientation of the bone core, will be rinsed with a cold 5% glucose solution to remove blood residues while maintaining the correct osmolarity (278 mOsm/L). Samples will then be fixed for 3 days in a 10% buffered formalin solution at pH 7.2 and then dehydrated in ascending series of alcohol rinses. After 5 days of preinfiltration in a 50% resin/alcohol solution, biopsies will be removed from the core drills and sample infiltration will be completed with methacrylate resin. After 12 days of polymerization, the samples will be cut along their longitudinal axis using a high-precision silicon carbide disc at 50 μm and then finished under running water with a series of polishing discs at approximately 30 ± 10 μm. They will then be mounted on slides and stained with acid fuchsin, toluidine blue and Von Kossa.

Following histological and histomorphometric analyses, the samples will be delivered to specialized and authorized companies for disposal, according to current legislation.

Statistical plan The statistical analysis will be performed by means of a computerized statistical package (SigmaStat 3.5, SPSS Inc., Germany). The data will be expressed as mean ± standard deviation and median (interquartile range), respectively, for parametric and non-parametric values.

Sample size calculation The aim of the study is to clinically compare different alveolar ridge preservation techniques.

Considering the outcomes of previously published studies, it was calculated that will be necessary to recruit 15 patients for each group to obtain a statistically significant result through a comparison between subpopulations with a statistical power of 95% and a significance of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years;
* Single-rooted tooth with indication for extraction and presenting adjacent teeth;
* Presence of type II defect;
* Sufficient bone height of the extraction site for the insertion of a standard implant (≥8.5 mm);
* Healthy oral mucosa with at least 3 mm of keratinized tissue;
* American Society of Anesthesiologists 3;
* Periodontal health or stability;
* Signature of informed consent.

Exclusion Criteria:

* Presence of general contraindications for oral surgery;
* Presence of inflammatory and autoimmune diseases;
* Uncontrolled diabetes (HbA1c 7%);
* History of tumors requiring chemotherapy or radiotherapy in the last 5 years;
* Previous therapy with bisphosphonates or high-dose corticosteroid therapy;
* Smoking (10 cigarettes/day);
* Allergy to bovine collagen;
* Pregnancy or breastfeeding;
* Lack of compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients needing for tooth extraction and possible implant insertion meeting inclusion and exclusion criteria were eligible
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-01-06 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
alveolar volume | 6 months post-extractive
  optical scanning comparison

SECONDARY OUTCOMES:
histomorphometric analysis | 6 months post-extraction
  bone volume/total volume

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Stacchi, Dr., Principal Investigator — University of Trieste, Department of Medicine, Surgery and Health Sciences
Locations (1):
- University of Trieste, Departmen of Medicine, Surgery, Health Sciences, Trieste, Trieste, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pramstraller M, Farina R, Simonelli A, Gotz W, Trombelli L. A Simplified Procedure for Biologically Oriented Alveolar Ridge Preservation: Clinical and Histological Findings From a Case Report. Clin Adv Periodontics. 2021 Dec;11(4):189-194. doi: 10.1002/cap.10120. Epub 2020 Sep 18. PMID 32945629
- [Background] Schwarz F, Obreja K, Mayer S, Ramanauskaite A, Sader R, Parvini P. Efficacy of autogenous tooth roots for a combined vertical and horizontal alveolar ridge augmentation and staged implant placement. A prospective controlled clinical study. J Clin Periodontol. 2022 May;49(5):496-505. doi: 10.1111/jcpe.13609. Epub 2022 Mar 8. PMID 35258131
- [Background] Araujo MG, Silva CO, Misawa M, Sukekava F. Alveolar socket healing: what can we learn? Periodontol 2000. 2015 Jun;68(1):122-34. doi: 10.1111/prd.12082. PMID 25867983